CLINICAL TRIAL: NCT06679790
Title: Trajectories of Change in Tourette Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021987
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Tourette Syndrome; Tic Disorders
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive Behavioral Intervention for Tics (CBIT) (Experimental): behavior therapy for tics
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics — All participants will receive 8 sessions of CBIT following a published treatment manual.

SUMMARY:
This K23 Career Development Award is designed to provide the training needed for the PI to achieve her long-term career goal of conducting independent, programmatic intervention research in developmental populations. The training will emphasize gaining expertise in higher-intensity, multi-method, within-subject data collection and analysis. This award builds on the PI's emerging experience in tic disorders and pediatric behavioral interventions, and her ability to quickly learn and apply advanced statistical methods. The award will extend the PI's training through the following short-term training goals: 1) multi-method data collection and integration (electronic momentary assessment [EMA], wearable devices, neurocognitive tasks), 2) leading and designing pediatric clinical trials, 3) managing and analyzing large, multilevel datasets, and 4) career development and contribution to the field. The PI has developed a training plan to accomplish these goals in concert with her mentors, a team of leading experts in the fields of psychiatry and psychology, who will closely monitor training through regular meetings. The highly structured training plan also includes a set of formal coursework and workshops for each training goal to complement the hands-on experience the PI will gain from leading the research project.

The objective of this proposal is to comprehensively map symptom change across time and during a behavioral intervention for youth with Persistent Tic Disorders (PTDs). PTDs affect approximately 1% of the population, can cause significant disability, have high rates of comorbidity, and are associated with a four-fold increase in suicide risk. Research has established that tic symptoms and their change over time are highly idiographic. However, first-line, evidence-based, existing interventions are "one-size-fits-all," and are only effective for 60% of patients. The current study aims to use advanced statistical methods and a novel theoretical framework to map the stability of tic patterns, along with systemic factors that relate to tic change over time. Study hypotheses, based on the literature and preliminary data, are that a) tic change patterns will be stable before intervention for all participants, b) disruption of stable patterns during the intervention phase will be associated with treatment response, and c) this disruption will depend on the specific driver of tic symptoms pre-intervention. N = 30 youth ages 12-17 with chronic tics will be recruited for the study. There will be three study phases: 1) pre-intervention (4 weeks), 2) intervention (8 weeks), and 3) post-intervention (4 weeks). Before and between each phase, participants will complete 4 traditional assessments to assess symptoms and treatment response. Throughout the 16 weeks of the study, we will collect EMA data focused on factors relevant to tics (4x per day), physiological data from wearable devices (passive, continuous), and neurocognitive task performance and tic video observation (1x per week). Results will inform efforts to develop individualized interventions for individuals with PTDs to improve treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of chronic motor and/or vocal tics, defined as tics for at least 1 year without a tic-free period of more than 3 consecutive months. Tics must not be due to a medical condition or the direct physiological effects of a substance.
2. At least moderate tic severity, defined as a Yale Global Tic Severity Scale44 total score ≥14 (≥9 for those with motor or vocal tics only).
3. Participants must be fluent in English to ensure comprehension of study measures and instructions.

Exclusion Criteria:

1. Previous diagnosis of psychosis or cognitive disability,
2. IQ < 80,
3. Substance abuse or dependence within the past year.
4. Current suicidal intent.
5. Changes in medication in the previous 4 weeks.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Clinical scales of tic change | 4 months
  ecological momentary assessment outcomes of tic change

CONTACTS AND LOCATIONS:
Overall Officials: Brianna Wellen, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States